CLINICAL TRIAL: NCT00506116
Title: Promoting Effective Recovery From Labor Urinary Incontinence: Prevention Reducing Birthing Risk
Brief Title: Promoting Effective Recovery From Labor Urinary Incontinence (PERL)
Acronym: PERL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01NR4007-9; R01NR004007 (NIH)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-05

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse; Perinatal Laceration; Second Stage Labor
Keywords: Pelvic floor muscle training; Self-directed pushing; Antenatal perineal massage
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse | interventions — Videotape Recording; Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Videotape, routine care, PME instruction — A 40 minute videotape about non-directed, spontaneous pushing and/or a videotape of antenatal perineal massage and pelvic muscle exerise (PME) at intake visit. The control women received routine care and PME instruction at intake visit.
Behavioral: PME practice and record keeping (in diaries)
Behavioral: Non-directed or directed,spontaneous or sustained pushing — Non-directed, spontaneous pushing (experimental group) with perineal massage vs. directed, sustained pushing during delivery.
Procedure: Data collection — Baseline at 20 weeks gestation; longitudinal at 35 weeks gestation, 6 weeks postpartum, 6 months postpartum, and 12 months postpartum

SUMMARY:
The purpose of this study is to determine whether pushing during labor that is controlled by the woman results in less birth-related injury and less postpartum urinary incontinence (UI).

DETAILED DESCRIPTION:
Birth related urinary incontinence (UI) is a predictor of UI in older women. Ways to protect the continence mechanism during delivery may diminish a woman's risk of UI later in life. We propose to study the functional anatomy of the pelvic floor as it relates to UI in women who are having their first baby. We hypothesize non-directed, spontaneous pushing is a protective strategy in decreasing the risk of immediate and long term UI. Longitudinal comparisons of pelvic floor characteristics will be taken at 35 week gestation and 6 weeks, 6 months, and 12 months postpartum. Study participants will be seen first at 20 weeks gestation for documentation of baseline levels of pelvic floor function, specifically voluntary and involuntary muscle strength, urinary continence status, and urethral support. They will be randomly assigned into non-directed, spontaneous (experimental) and directed, sustained pushing (control) groups. Alterations that may occur in urethral support before and after birth will be described through non-invasive urethral ultrasound.

ELIGIBILITY:
Inclusion Criteria:

Women giving birth for the first time who are:

1. Age 18 years or older
2. Less than 20 weeks gestation
3. Expected vaginal birth without use of epidural analgesia
4. Plan to reside in Southeast Michigan for one year following the birth of the infant.

Exclusion Criteria:

1. History of genito-urinary or neuro-muscular pathology
2. Previous pregnancy carried beyond 20 weeks gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 1996-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Leakage Index ( | 20 and 35 weeks gestation, and 6 weeks, 6 months, and 12 months postpartum

SECONDARY OUTCOMES:
Perineal status (Digital, speculum, chart review, ultrasound) | 35 week gestation and 6 weeks, 6 months, and 12 months postpartum
Pelvic Organ Prolapse Quantification System (POPQ) | 35 weeks gestation and 6 weeks, 6 months, and 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn M Sampselle, PhD,RNC,FAAN, Principal Investigator — University of Michgan School of Nursing
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] DeLancey JO, Sampselle CM, Punch MR. Kegel dyspareunia: levator ani myalgia caused by overexertion. Obstet Gynecol. 1993 Oct;82(4 Pt 2 Suppl):658-9. PMID 8378003
- [Result] Sampselle CM, Miller JM, Luecha Y, Fischer K, Rosten L. Provider support of spontaneous pushing during the second stage of labor. J Obstet Gynecol Neonatal Nurs. 2005 Nov-Dec;34(6):695-702. doi: 10.1177/0884217505281904. PMID 16282227
- [Result] Antonakos CL, Miller JM, Sampselle CM. Indices for studying urinary incontinence and levator ani function in primiparous women. J Clin Nurs. 2003 Jul;12(4):554-61. doi: 10.1046/j.1365-2702.2003.00747.x. PMID 12790869
- [Result] Armstrong SM, Miller JM, Benson K, Jain S, Panagopoulos K, DeLancey JO, Sampselle CM. Revisiting reliability of quantified perineal ultrasound: Bland and Altman analysis of a new protocol for the rectangular coordinate method. Neurourol Urodyn. 2006;25(7):731-8. doi: 10.1002/nau.20299. PMID 16897749
- [Result] Roberts JM, Gonzalez CBP, Sampselle C. Why do supportive birth attendants become directive of maternal bearing-down efforts in second-stage labor? J Midwifery Womens Health. 2007 Mar-Apr;52(2):134-141. doi: 10.1016/j.jmwh.2006.11.005. PMID 17336819